CLINICAL TRIAL: NCT04754841
Title: SURVIVAL AND FUNCTIONALITY EVALUATION IN VITRO IN CRYOPRESERVED PLATELETS
Brief Title: STUDY OF SURVIVAL AND FUNCTIONALITY IN CRYOPRESERVED PLATELETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HOSPITAL BRITANICO DE BUENOS AIRES (Other)
Responsible Party: Principal Investigator, JHON ALEXANDER AVILA RUEDA, Specialist in Internal Medicine an Hematology, HOSPITAL BRITANICO DE BUENOS AIRES
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1021
Record Dates: First submitted 2021-02-07; First posted 2021-02-15 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Platelet Cryopreservation; Platelet Survival
Keywords: SURVIVAL; FUNCTIONALITY; CRYOPRESERVED PLATELETS; IN VITRO

STUDY DESIGN:
Intervention Model Description: A blind experimental study will be carried out (those who evaluate viability and functionality of platelets will not know the cryopreservation times or the concentration of the cryopreservative)
  Aliquots of platelets with group and factor A +, A-, B +, B-, AB +, AB-, O + and O- obtained from those people who come to the hemotherapy center as voluntary donors and who in turn express their decision to participate in this protocol by signing an informed consent designed for this purpose.
Masking Description: Cryopreserved samples will be labeled with a code unknown to the researcher and those who process the sample in the laboratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SURVIVAL AND FUNCTIONALITY INVITRO IN CRYOPRESERVED PLATELETS (Experimental): Platelet concentrates will be administered 3 alternatives of cryopreservative solution: 5% dimethylsulfoxide (solution 1), 5% dimethylsulfoxide plus 160 mg of 5% dextrose (solution 2) and 5% dimethylsulfoxide plus 2% albumine (solution 3 ). They will then be frozen at -80 ° C and their survival and functionality will be subsequently evaluated in vitro.
  Interventions: Other: platelet cryopreservation

INTERVENTIONS:
Other: platelet cryopreservation — The cryopreservation of platelets will be carried out using as alternatives of cryopreservative solution: 5% dimethylsulfoxide alone (solution 1) or combined with 5% dextrose 160 mg (solution 2) or with 2% albumin (solution 3) and then be frozen at -80 ° C

SUMMARY:
Platelets correspond to one of the most widely used blood components in transfusion medicine, given their importance in the prevention of bleeding disorders in patients with multifactorial thrombocytopenia and non-immunological etiology, as well as in the management of traumatic or blood-related bleeding. surgical treatments. Given its wide margin of use and the constant demand for it for use within the different management schemes and procedures associated with the medical act, it is the objective of both hemotherapy services and blood banks and blood products to have availability component constant to meet such requirements. The main problem of this resource is its short useful life (5 to 7 days) which limits its availability, especially in the Latin American context where the production of blood components as well as the resources allocated for this purpose by state entities to blood banks are generally limited. Cryopreservation at -80 ° C using Dimethylsulfoxide as a preservative solution is a technique used since the 1950s to prolong platelet survival, the improvement of which has been remarkable in recent years, thus constituting an alternative for the resolution of this problem.

DETAILED DESCRIPTION:
HYPOTHESIS: Through cryopreservation it is possible to prolong the survival time of platelets up to 4 times, compared to those preserved under the conventional method, maintaining a viability equal to or greater than 50%.

There is a direct relationship between survival time, viability and functionality of cryopreserved platelets depending on the model of cryoprotective solution used.

PRIMARY OUTCOME: survival of cryopreserved platelets greater than 28 days SECUNDARY OUTCOME: viability of cryopreserved platelets greater than 50%

INCLUSION CRITERIA: Concentrates from donors over 18 years of age who meet the requirements established by law 22990 (Of Argentine Republic) for donating blood and blood components will be included in this study, from whom a number of platelets greater than or equal to 3 x10 E11 can be collected.

EXCLUSION CRITERIA: Platelet concentrates that present any of the following characteristics will be excluded from the investigation:

Concentrates that have not met all of the standards required for use in humans or that at the time of the study more than 24 hours have passed since they were obtained.

A blind experimental study will be carried out (those who evaluate viability and functionality of platelets will not know the cryopreservation times or the concentration of the cryopreservative)

Aliquots of platelets with group and factor A +, A-, B +, B-, AB +, AB-, O + and O- obtained from those people who come to the hemotherapy center as voluntary donors and who in turn express their decision to participate in this protocol by signing an informed consent designed for this purpose. Obtaining platelets will be performed by apheresis using the Trima ACCEL cell separator, version 7.0, TERUMO BCT brand.

A minimum total of 3.3 x1011 platelets will be obtained in a volume between 200 - 300 ml, for each donor.

Group A: It will consist of 70 aliquots of 3 ml each with 1.9 x109 platelets to which a solution composed of: 1 ml obtained from the following mixture will be added (0.8 ml of 100% Dimethylsulfoxide (DMSO) and 4 ml of 0 sodium chloride , 9%). They will then be frozen at -80 ° C.

B Group: It will be made up of 70 aliquots of 3 ml each with 1.9 x109 platelets to which will be added a solution composed of: 0.4 ml of 20% UNC brand albumin and 0.6 ml obtained from the following mixture (1.4 ml of Dimethylsulfoxide (DMSO) 100% and 4 ml of Dextrose 5%). They will then be frozen at -80 ° C.

Group C: It will be made up of 70 aliquots of 3 ml each with 1.9 x109 platelets to which will be added a solution composed of: 0.4 ml of 20% UNC brand albumin and 0.6 ml obtained from the following mixture (1.4 ml of Dimethylsulfoxide (DMSO) 100% and 4 ml of 0.9% sodium chloride). They will then be frozen at -80 ° C.

A group of 71 aliquots of 3 ml each with 1.9 x109 irradiated platelets kept at 22 ° C under constant stirring for 5 days (twenty-four aliquots for each period of time evaluated) will be used as a reference for the comparison of results (group N).

Viability:

It will be evaluated through the platelet count carried out by the Beckman-Coulter system, the measurement of the pH of the cryopreserved platelets after being thawed (expected values between 6.4 and 7.4) and the immunophenotyping of the platelets by flow cytometry (CMF) using fluorescent anti CD61-PE antibodies.

Functionality:

It will be evaluated from the immunophenotyping of platelets by flow cytometry (CMF) using fluorescent anti-CD41 and anti-CD62-FITC antibodies.

Before carrying out the CMF analysis, 4 microliters of a 50 mmol ADP solution will be added to each sample in order to induce platelet activation.

Both the viability analysis and the functionality of the cryopreserved product will be carried out by 3 biochemists, collaborating members of the research in the biochemical analysis laboratory of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Concentrates from donors over 18 years of age who meet the requirements established by law 22990 for donating blood and blood components will be included in this study, from whom a number of platelets greater than or equal to 3 x10 E11 can be collected

Exclusion Criteria:

* Platelet concentrates that present any of the following characteristics will be excluded from the investigation:

Concentrates that have not met all of the standards required for use in humans or that at the time of the study more than 24 hours have passed since they were obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-08-28 (Estimated); Study Completion 2022-02-02 (Estimated)

PRIMARY OUTCOMES:
survival of cryopreserved platelets greater than 28 days | Between 1 and 3 months

SECONDARY OUTCOMES:
viability of cryopreserved platelets greater than 50% | Between 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GLENDA ERNST, Study Chair — HOSPITAL BRITANICO DE BUENOS AIRES; JHON AVILA, Principal Investigator — HOSPITAL BRITANICO DE BUENOS AIRES
Locations (2):
- Argentina (2):
  - Hospital Britanico Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson L, Cameron M, Waters L, Padula MP, Marks DC. The impact of refrigerated storage of UVC pathogen inactivated platelet concentrates on in vitro platelet quality parameters. Vox Sang. 2019 Jan;114(1):47-56. doi: 10.1111/vox.12730. Epub 2018 Nov 30. PMID 30499111
- [Result] 7. Bohonek, Milos;Cryopreservation of Platelets: Advances and Current Practice; Cryopreservation Biotechnology in Biomedical Sciences ;2018;Chapter4;P47-66
- [Result] Waters L, Cameron M, Padula MP, Marks DC, Johnson L. Refrigeration, cryopreservation and pathogen inactivation: an updated perspective on platelet storage conditions. Vox Sang. 2018 May;113(4):317-328. doi: 10.1111/vox.12640. Epub 2018 Feb 14. PMID 29441601
- [Result] Eker I, Yilmaz S, Cetinkaya RA, Pekel A, Unlu A, Gursel O, Yilmaz S, Avcu F, Musabak U, Pekoglu A, Ertas Z, Acikel C, Zeybek N, Kurekci AE, Avci IY. Generation of Platelet Microparticles after Cryopreservation of Apheresis Platelet Concentrates Contributes to Hemostatic Activity. Turk J Haematol. 2017 Mar 1;34(1):64-71. doi: 10.4274/tjh.2016.0049. Epub 2016 Apr 18. PMID 27094612